CLINICAL TRIAL: NCT01069341
Title: Ranibizumab in Subjects With Dense Cataract and Rubeosis Due to Proliferative Diabetic Retinopathy (PDR)
Brief Title: Use of Ranibizumab to Treat Rubeosis in Diabetics Prior to Cataract Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bhagat, Neelakshi, M.D., M.P.H. (Individual)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF 4297s
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Rubeosis Iridis; Proliferative Diabetic Retinopathy
Keywords: Rubeosis; Neovascularization of iris; Proliferative diabetic retinopathy; PDR; Cataract
MeSH Terms: conditions — Cataract | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): All subjects enrolled received treatment with identical dosage of Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreally administered 0.5mg ranibizumab, 3 doses administered monthly.
  Other Names: Lucentis

SUMMARY:
The purpose of this study was to determine the safety of ranibizumab: a) as a surgical adjunct during cataract surgery in subjects with proliferative diabetic retinopathy (PDR) induced rubeosis and, b) in treatment of proliferative diabetic retinopathy (PDR).

DETAILED DESCRIPTION:
This is an open-label, Phase I study of intravitreally administered 0.5mg ranibizumab in diabetic subjects presenting initially with dense cataract and proliferative diabetic retinopathy induced rubeosis. Ten subjects will be enrolled at a single center over a 10 month period. Patients will be followed for a total of 12 months in the treatment phase and will have safety follow-ups at Months 18 and 24. Eligibility for study entry will be determined by the principal investigator.

Consented, enrolled subjects will receive multiple open-label intravitreal injections of 0.5 mg ranibizumab administered every month for 3 doses (loading dose on Day 0 and at Months 1 and 2) followed by as needed re-treatment based on specified criteria for the remainder of the study period. Subjects can receive a maximum of eight injections of ranibizumab during the study. All subjects will undergo cataract surgery after the first ranibizumab injection. Only one eye will be designated as the study eye for the duration of the study to receive the ranibizumab injections.

All subjects will be evaluated with best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity, intraocular pressure measurement, ophthalmological examination, slit lamp photography, gonioscopy, fundus photography, fundus fluorescein angiography and Optical Coherence Tomography (OCT). An ultrasound will be done as needed. Best corrected ETDRS visual acuity and intraocular pressure measurements will be performed on both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Subjects with diabetes mellitus
* Subjects with proliferative diabetic retinopathy induced rubeosis
* Be willing to undergo cataract surgery
* HgbA1c level < 12%

Exclusion Criteria:

* History of glaucoma surgery
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis
* Intraocular surgery in the study eye within 60 days preceding Day 0
* History of prior pars plana vitrectomy in the study eye
* Positive pregnancy test
* HbA1c >12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neelakshi Bhagat, MD, MPH, Principal Investigator — NJMS / UMDNJ
Locations (1):
- Njms / Umdnj, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the patients seen in the Ophthalmology Department at the University of Medicine and Dentistry of New Jersey.
Groups:
- All Subjects With Treatment: All subjects received o.5 mg of ranibizumab injections monthly for 3 months
Period: Overall Study
Arm/Group | All Subjects With Treatment
Started | 4
Completed | 3
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects With Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event (AE)
Description: Incidence and severity of AEs that were cataract surgery related (for instance, hyphema and vitreous hemorrhage) and AEs that occurred during the treatment of proliferative diabetic retinopathy (PDR).
Time Frame: first 12 months
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Number; unit: participants
Groups:
- All Subjects: 0.5 mg ranibizumab, intravitreal injection
Arm/Group | All Subjects
Number analyzed (Participants) | 4
participants | 0

2. Secondary Outcome: Presence of Neovascularization of Iris (NVI) or Neovascularization of the Angle (NVA)
Description: Presence of neovascularization of iris (NVI) or neovascularization of the angle (NVA) as assessed by gonioscopy at months 3, 7 and 12
Time Frame: months 3, 7 and 12
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 4
participants
  Month 3 | 0
  Month 7 | 0
  Month 12 | 0

3. Secondary Outcome: Presence of Proliferative Diabetic Retinopathy (PDR)
Description: Presence of proliferative diabetic retinopathy by fluorescein angiogram
Time Frame: at month-12
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 4
participants | 0

4. Secondary Outcome: Macular Volume
Description: Macular volume (millimeters cubed [mm3]) by Stratus OCT
Time Frame: at months-1,3,7, and 12
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Mean (Standard Deviation); unit: Macular volume (millimeters cubed)
Arm/Group | All Subjects
Number analyzed (Participants) | 4
Macular volume (millimeters cubed)
  Month 1 | 7.47 (1.00)
  Month 3 | 6.94 (0.57)
  Month 7 | 6.40 (0.61)
  Month 12 | 6.64 (0.25)

5. Secondary Outcome: Mean Time to Re-treatment
Description: Mean time to re-treatment following the initial three monthly loading doses of ranibizumab (months)
Time Frame: first 12 months
Population: All subjects' data was included
Measure: Mean (Standard Deviation); unit: months
Arm/Group | All Subjects
Number analyzed (Participants) | 4
months | 1 (0.73)

6. Secondary Outcome: Mean Number of Ranibizumab Injections
Description: Mean number of ranibizumab injections required through month 12
Time Frame: first 12 months
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Mean (Standard Deviation); unit: Number injections
Arm/Group | All Subjects
Number analyzed (Participants) | 4
Number injections | 3.5 (1.0)

7. Secondary Outcome: Mean Number of PRP Laser Treatments
Description: Mean number of PRP laser treatments required through month 12
Time Frame: first 12 months
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Mean (Standard Deviation); unit: PRP Laser treatments
Arm/Group | All Subjects
Number analyzed (Participants) | 4
PRP Laser treatments | 0.5 (1.0)

8. Secondary Outcome: Mean Change in Intraocular Pressure (IOP)
Description: Mean change in IOP (mm Hg) from baseline to months-3, 7, and 12.
Time Frame: at months-3,7, and 12
Population: All subjects' data was analyzed, no subjects were excluded
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Subjects
Number analyzed (Participants) | 4
mmHg
  from baseline to month-3 | 0 (1.63)
  from baseline to month-7 | 1 (4)
  from baseline to month-12 | 0 (5.57)

ADVERSE EVENTS:
Time Frame: Day 1 to Month-24
Arm/Group | All Subjects With Treatment
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | All Subjects With Treatment (N=4)
Foot amputation surgery pre-scheduled prior to enrollment (Musculoskeletal and connective tissue disorders) | 1/1 (1) — Hospitalization for a diabetic foot ulcer with a foot amputation scheduled prior to enrollment, 24 days after 1st injection.
Hospitalization for congestive heart failure attributed to uncontrolled diabetes (Cardiac disorders) | 1/1 (1) — 2 months after 4th injection; 3 months after 4th injection: hospitalizations for CHF attributed to uncontrolled diabetes
Hospitalization for hyperkalemia and CHF, attributed to renal insufficiency (Cardiac disorders) | 1/1 (1) — 2 months after 5th injection: hospitalization for hyperkalemia and CHF, attributed to renal insufficiency due to uncontrolled diabetes
Hospitalization for exacerbation of CHF (Cardiac disorders) | 1/1 (1) — 4 months after 5th injection: hospitalization for exacerbation of CHF
Hospitalization for pleural effusion, CHF, and worsening of pre-existing foot ulcers (MRSA) (Cardiac disorders) | 1/1 (1) — 5 months after 5th injection: hospitalization for pleural effusion, CHF and worsening of pre-existing bilateral foot ulcers which cultures identified as MRSA
Hospitalization for chronic osteomyelitis (Musculoskeletal and connective tissue disorders) | 1/1 (1) — 14 months after 5th injection: hospitalization for chronic osteomyelitis
Hospitalization for congestive heart failure and renal insufficiency (Renal and urinary disorders) | 1/1 (1) — 9 months after 3rd injection
Hospitalization for flare-up of pre-existing gastritis (Gastrointestinal disorders) | 1/1 (1) — 15 months after 3rd injection: hospitalization for flare-up of pre-existing gastritis

LIMITATIONS AND CAVEATS:
Uncontrolled pilot study with a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No